CLINICAL TRIAL: NCT03352661
Title: Influence of an Endometrioma on Oocyte Quality
Acronym: ENDOVOC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: IVI Vigo (Other)
Responsible Party: Sponsor
Other Study IDs: 1311-VGO-137-EM
Record Dates: First submitted 2017-01-17; First posted 2017-11-24 (Actual); Last update posted 2017-11-24 (Actual); Status verified 2017-01

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Endometriosis: No drugs are administered. It is an observational study. Collect retrospectively data
  Interventions: Other: Collect retrospectively data
- No endometriosis: No drugs are administered. It is an observational study. Collect retrospectively data
  Interventions: Other: Collect retrospectively data

INTERVENTIONS:
Other: Collect retrospectively data — Collect retrospectively data

SUMMARY:
The purpose of this study is to evaluate if there are differences in oocyte quality depending on whether these oocytes come from an ovary in contact with an endometrioma.

DETAILED DESCRIPTION:
There is no consensus for whether an endometrioma influences oocyte quality, as well as the possible mechanisms that induce them.

In this study, the oocyte maturation will proof oocyte quality: This mean, the percentage of oocytes in metaphase II obtained after stimulation, as well as the rate of oocytes fertilized in direct contact with an endometrioma.

ELIGIBILITY:
Inclusion Criteria:

* Patients <40 years, BMI <30kg / m2,

Exclusion Criteria:

-

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients <40 years, BMI <30kg / m2,
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-01; Primary Completion 2017-11 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of mature oocytes | Up to 36 months
  Number of MII oocytes from the total of cumulus granulosa cell-oocyte complex by 100
Fertilization rate | Up to 36 months
  Number of oocytes with pronuclear activation after ICSI procedure from the total oocytes microinjected by 100

CONTACTS AND LOCATIONS:
Overall Officials: Elkin Muñoz, Principal Investigator, Principal Investigator — IVI Vigo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Garcia-Velasco JA, Mahutte NG, Corona J, Zuniga V, Giles J, Arici A, Pellicer A. Removal of endometriomas before in vitro fertilization does not improve fertility outcomes: a matched, case-control study. Fertil Steril. 2004 May;81(5):1194-7. doi: 10.1016/j.fertnstert.2003.04.006. PMID 15136074
- [Background] Garrido N, Navarro J, Remohi J, Simon C, Pellicer A. Follicular hormonal environment and embryo quality in women with endometriosis. Hum Reprod Update. 2000 Jan-Feb;6(1):67-74. doi: 10.1093/humupd/6.1.67. PMID 10711831
- [Background] Filippi F, Benaglia L, Paffoni A, Restelli L, Vercellini P, Somigliana E, Fedele L. Ovarian endometriomas and oocyte quality: insights from in vitro fertilization cycles. Fertil Steril. 2014 Apr;101(4):988-93.e1. doi: 10.1016/j.fertnstert.2014.01.008. Epub 2014 Mar 3. PMID 24602751